CLINICAL TRIAL: NCT02236403
Title: Diagnosis of Demodex Blapharitis and Treatment With Ivermectin Gel 0.1%/ Metronidazole 1%
Brief Title: Treatment of Demodex Blepharitis With Ivermectin Gel 0.1% Plus Metronidazole 1%
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Universidad Nacional de Colombia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: demodex0.1
Record Dates: First submitted 2014-09-08; First posted 2014-09-10 (Estimated); Last update posted 2021-05-06 (Actual); Status verified 2021-05

CONDITIONS: Chronic Blepharitis
Keywords: Blepharitis , Demodex, Ivermectin, Metronidazole
MeSH Terms: conditions — Blepharitis | interventions — Ivermectin; 22,23-dihydroavermectin B(1)a; avermectin H2B1b

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ivermectin 0.1% Metronidazole 1% (Experimental): 30 patients will receive the treatment and at 15 days a second visit will be done and changes in mite counts will be determinated and correlated with symtoms and signs.
  Interventions: Drug: Ivermectin 0.1% Metronidazole 1%
- Control (Placebo Comparator): 30 volunters with no signs of blepharitis and with eyelashes with no demodex .None intervention. Symptoms and signs will be compared with experimental group
  Interventions: Other: None intervention

INTERVENTIONS:
Drug: Ivermectin 0.1% Metronidazole 1%
  Other Names: 22,23-dihydroavermectin B1a + 22,23-dihydroavermectin B1b
  Arms: Ivermectin 0.1% Metronidazole 1%
Other: None intervention — Volunteers with no signs of blepharitis and with eyelashes with no demodex. Symptoms and signs will be compared with experimental group
  Arms: Control

SUMMARY:
Blepharitis is a endemic inflammatory disease caused mainly by Demodex folliculorum and Demodex Brevis, This mites are often associated with anaerobic bacteria that produces a skin inflammation, so a intervention that reduces the number of mites and bacteria would be desirable. Ivermectin a macrolid compound have demonstrated activity against scabies and lice in humans and in animals and a single application have show a good response in lice eradication.

In this study , investigators will determinate the security and effectiveness of this compound in the eradication of mites

ELIGIBILITY:
Inclusion Criteria:

* • Patients with symptomatic Demodex blepharitis for duration of at least 3 months.

  * Age range: 18 yeras and older.
  * Both genders and all ethnic groups comparable with the local community.
  * Able to understand and willing to sign a written informed consent
  * Able and willing to cooperate with the investigational plan.
  * Able and willing to complete all mandatory follow-up visits.

Exclusion Criteria:

* • Patients who are currently engaged in another clinical trial, unwilling or unable to give consent, to accept randomization, or to return for scheduled visits.

  * Children under 18.
  * Pregnant women or expecting to be pregnant during the study.
  * Systemic immune deficient conditions such as AIDS or under systemic immunosuppressant.
  * Concomitant use of ophthalmic topical medications (excluding non-preserved tear substitutes).
  * Concomitant use of systemic antibiotics or steroids.
  * Contact lens wear
  * Active ocular infection or allergy
  * Unable to close eyes or uncontrolled blinking Previous allergic reaction to metronidazole and / or ivermectin

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2014-10; Primary Completion 2015-01 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Erradication of Demodex mites | 2 months
  Reduction in mites count after treatment compared to baseline data. If mites are not observed in the last visit a complete eradication will be considered. Patients with one or more mites will be considered as a incomplete eradication

SECONDARY OUTCOMES:
Change in lid margin rednes and bulbar conjunctival hyperemia categorized from 0 (none) to 3 (severe) according to the next score | 2 months
  Change in lid margin rednes and bulbar conjunctival hyperemia categorized from 0 (none) to 3 (severe) according to the next score
  * None (0) = normal
  * Mild (1) = Slight localized injection
  * Moderate (2) = pink color
  * Severe (3) = dark redness

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Engativa, Bogotá, Colombia